CLINICAL TRIAL: NCT01729364
Title: Colloid vs Crystalloid Infusion Postoperative in CABG Patients Regarding Renal Hemodynamics and Function
Brief Title: Fluid Investigation Colloid vs Crystalloid Reg. Renal Hemodynamics and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jenny Skytte Larsson, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: vätskestudien
Record Dates: First submitted 2012-11-09; First posted 2012-11-20 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Renal Impairment
Keywords: elective CABG; renal impairment; GFR; renal blood flow; colloid; crystalloid; thermodilution technique; oxygen supply demand
MeSH Terms: conditions — Renal Insufficiency | interventions — Crystalloid Solutions; Ringer's Lactate; Colloids; HES 130-0.4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- crystalloid (Experimental): crystalloid fluid administration, Ringer-acetat 20ml/kg under 30 minutes
  Interventions: Drug: crystalloid
- colloid (Experimental): colloidal fluids administration, HES 6% (130/0,4) 7ml/kg under 30 minutes
  Interventions: Drug: colloid

INTERVENTIONS:
Drug: crystalloid
  Other Names: Ringer Lactate; NaCl
  Arms: crystalloid
Drug: colloid
  Other Names: Voluven; Venofundin; Tetraspan
  Arms: colloid

SUMMARY:
Comparing the effects of crystalloid versus colloid fluid resuscitation in CABG patients postoperatively regarding renal blood flow, glomerular filtration rate and renal oxygen demand.

DETAILED DESCRIPTION:
Due to blood loss and SIRS postoperative hypovolemia is a usual feature after CABG surgery. Substantial controversy persists regarding the best choice of fluid to be used for resuscitation in this setting regarding renal function and oxygen supply-demand matching. In our study we aim to investigate differences in functional renal parameters by dividing patients postoperatively in two groups, substituted either with crystalloid fluid, Ringer-Acetat, 20 ml/kg or colloid, HES 6% (130/0,4) 10 ml/kg under 20 minutes. Central and renal hemodynamics will be measured before (baseline) and after fluid administration by blood sampling and thermodilution in both pulmonary artery catheter and renal vein catheter. Measurement endpoints will mainly consist of central hemodynamics, renal blood flow, GFR and renal oxygen extraction rate which we aim to compare between groups.

ELIGIBILITY:
Inclusion Criteria:

* elective fast track CABG patients, postoperative

Exclusion Criteria:

* hemodynamic instability
* preoperative renal impairment
* major postoperative bleeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline and differences inbetween groups in glomerular filtration rate, measured at different timepoints | 125min after baseline-measures
  GFR measured by thermodilution and blood- and urine sampling baseline1 (0min), baseline2 (+30min), timepoint1 (+65min), tp2 (+85min), tp3 (+105min), tp4 (+125min)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Skytte Larsson, MD, Principal Investigator — Sahlgrenska University Hospital; Sven-Erik Ricksten, Professor, Study Chair — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital/Thoracic Intensive Care, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Derived] Skytte Larsson J, Bragadottir G, Krumbholz V, Redfors B, Sellgren J, Ricksten SE. Effects of acute plasma volume expansion on renal perfusion, filtration, and oxygenation after cardiac surgery: a randomized study on crystalloid vs colloid. Br J Anaesth. 2015 Nov;115(5):736-42. doi: 10.1093/bja/aev346. PMID 26475802